CLINICAL TRIAL: NCT00266760
Title: Episodic Ataxia Syndrome: Genotype-phenotype Correlation and Longitudinal Study
Brief Title: Characteristics of Episodic Ataxia Syndrome
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: RDCRN 5302; U54RR019482-03 (NIH)
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Episodic Ataxia Syndrome; Cerebellar Diseases
MeSH Terms: conditions — Episodic Ataxia; Cerebellar Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood

SUMMARY:
Episodic ataxia (EA) is a rare genetic disease characterized by episodes of imbalance, incoordination, and slurring of speech. The underlying cause of EA is only partly understood, and currently there are no established treatments. There is also little information about the link between EA's clinical features and its genetic basis. The purpose of this study is to better characterize EA and disease progression. In turn, this may direct the development of future treatments.

DETAILED DESCRIPTION:
Attacks of ataxia, or the loss of ability to coordinate muscular movement, are often triggered by stress or exertion. EA is likely caused by an inherited genetic mutation; many individuals with EA have abnormalities in the KCNA1 or CACNA1A genes. To date, two known subtypes of EA have been identified, and other types likely exist. Specific characteristics of each EA subtype, however, have not been adequately described. The purpose of this study is to better define the clinical features and genetic basis of the various subtypes of EA and to evaluate disease progression. The study will also establish relevant study endpoints for use in future therapeutic trials.

This multi-center observational study will involve both a cross-sectional data analysis and a prospective longitudinal analysis. Participants will initially attend an outpatient study visit that will last 7 hours. This initial evaluation will include a medical history, a physical examination, neurological testing, and an ataxia assessment. Blood will be collected for genetic testing. Additionally, the following procedures may be conducted: ocular motor test, electromyography/nerve conduction study, electroencephalogram, MRI, and digital videotaping. Follow-up evaluations will occur on a yearly basis for at least 2 years; each will last 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* A clinically confirmed diagnosis of episodic ataxia as defined by one of the following three features:

  1. Clear-cut episodes of recurrent, transient ataxia
  2. Mutation confirmed in KCNA1 or CACNA1A
  3. Ataxic features with a first degree relative with episodic ataxia

Exclusion Criteria:

* Any other disorder known to cause episodic ataxia

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with episodic ataxia
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2006-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W. Baloh, MD, Study Chair — University of California, Los Angeles; Joanna C. Jen, MD, PhD, Principal Investigator — University of California, Los Angeles; Tracey Graves, MD, Principal Investigator — Institute of Neurology and National Hospital for Neurology; Yoon-Hee Cha, MD, Principal Investigator — University of California, Los Angeles
Locations (6):
- United States (4):
  - Reed Neurological Research Center, UCLA, Los Angeles, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Rochester School of Medicine, Rochester, New York
- London Health Sciences Centre, London, Ontario, Canada
- Institute of Neurology, Center for Neuromuscular Disease, Queen Square, London, United Kingdom

REFERENCES:
- [Background] Jen J, Kim GW, Baloh RW. Clinical spectrum of episodic ataxia type 2. Neurology. 2004 Jan 13;62(1):17-22. doi: 10.1212/01.wnl.0000101675.61074.50. PMID 14718690
- [Background] Sasaki O, Jen JC, Baloh RW, Kim GW, Isawa M, Usami S. Neurotological findings in a family with episodic ataxia. J Neurol. 2003 Mar;250(3):373-5. doi: 10.1007/s00415-003-0994-3. No abstract available. PMID 12749331
- [Background] Denier C, Ducros A, Vahedi K, Joutel A, Thierry P, Ritz A, Castelnovo G, Deonna T, Gerard P, Devoize JL, Gayou A, Perrouty B, Soisson T, Autret A, Warter JM, Vighetto A, Van Bogaert P, Alamowitch S, Roullet E, Tournier-Lasserve E. High prevalence of CACNA1A truncations and broader clinical spectrum in episodic ataxia type 2. Neurology. 1999 Jun 10;52(9):1816-21. doi: 10.1212/wnl.52.9.1816. PMID 10371528
- [Result] Graves TD, Cha YH, Hahn AF, Barohn R, Salajegheh MK, Griggs RC, Bundy BN, Jen JC, Baloh RW, Hanna MG; CINCH Investigators. Episodic ataxia type 1: clinical characterization, quality of life and genotype-phenotype correlation. Brain. 2014 Apr;137(Pt 4):1009-18. doi: 10.1093/brain/awu012. Epub 2014 Feb 26. PMID 24578548